CLINICAL TRIAL: NCT04332627
Title: Comparison of Quality of Recovery Score (QoR-15) According to Neuromuscular Blocking Reversal Agent in Laparoscopic Cholecystectomy: Sugammadex vs. Neostigmine
Brief Title: Comparison of QoR-15 in Laparoscopic Cholecystectomy: Sugammadex vs. Neostigmine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, JiWon Han, clinical instructor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: B-1910/571-004
Record Dates: First submitted 2020-04-01; First posted 2020-04-02 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Neuromuscular Blockade Reversal Agent; Sugammadex; Neostigmine; Quality of Recovery; Laparoscopic Cholecystectomy
MeSH Terms: interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sugammadex (Active Comparator): sugammadex 2mg/kg or 4mg/kg according to Train-of-four count (TOF 0 : 4mg/kg, TOF 1-4 : 2mg/kg)
  Interventions: Drug: Sugammadex
- neostigmine (Placebo Comparator): with glycopyrrolate 0.4mg, neostigmine 0.02mg/kg or 0.04mg/kg or 0.05mg/kg according to Train-of-four count (TOF 0 : wait until TOF 2, TOF2-3: 0.05mg/kg, TOF4: 0.04mg/kg)
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Sugammadex — sugammadex 2mg/kg or 4mg/kg according to Train-of-four count (TOF 0 : 4mg/kg, TOF 1-4 : 2mg/kg)
  Arms: sugammadex
Drug: Neostigmine — with glycopyrrolate 0.4mg, neostigmine 0.02mg/kg or 0.04mg/kg or 0.05mg/kg according to Train-of-four count (TOF 0 : wait until TOF 2, TOF2-3: 0.05mg/kg, TOF4: 0.04mg/kg)
  Arms: neostigmine

SUMMARY:
The quality of recovery in patients who were reversed neuromuscular blockade by using Sumamadex and Neostigmine in laparoscopic cholecystectomy was compared through the QoR(Quality of Recovery)-15 questionnaire.

DETAILED DESCRIPTION:
Quality of Recovery questionnaire includes five details (Emotional status, Physical comfort, Physiological support, Physical independece, Pain), and is a proven method of reliability, consistency and validity for evaluating recovery from surgery and anesthesia.

After laparoscopic cholecystectomy, patients experience various discomforts such as pain, nausea, vomiting, and placebo due to general anesthesia.

Neostigmine has side effects such as crampy abdominal pain, nausea and vomiting. In addition, residual neuromuscular blockade was higher in neostigmine compared with sugammadex.

Although sugammadex expected to improve patient's recovery, it is still controversial that sugammadex contributes to clinically meaningfull difference compared with neostigmine.

Therefore, the aim of our study is comparison of quality of recovery through QoR-15 questionnaire in patients who were reversed neuromuscular blockade by using sugammadex and neostigmine in laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent laparoscopic cholecystectomy aged 20-70

Exclusion Criteria:

* neuromuscular disease
* allergy to rocuronium, sugammadex, neostigmine
* cognitive impairment ( disable to answer the questionnaire )
* refuse to participate

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2020-05-21 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery(QoR)-15 questionnaire score | preoperative 1 days to postoperative 2 days
  the difference of Quality of Recovery(QoR)-15 score between preoperative and postoperative 1 and 2 days (minimum value : 0, maximum value : 150, the higher the score, the better the result)

SECONDARY OUTCOMES:
recovery time | perioperative - until 48hours
  from injection of sugammadex or neostigmien to extubation and confirm of adequate spontaneous breathing
PACU(post-anesthesia care unit) stay time | perioperative - until 48hours
  from entry of PACU to go general ward
postoperative pain score | at postoperative 30minutes, 6hours, 24hours
  postoperative pain score measured by 11-point NRS(numerical rating scale) score (minimum : 0, maximum : 11, the lower the score, the lesser pain)
the incidence of administration of postoperative rescue drug | perioperative - until 72hours
  administration of analgesic drug and anti-emetic drug for postoperative management
hospital stay | preoperative - until discharge (usually 48 hours to 72hours)
  days of hospital stay
urinary retention | postoperative - until discharge (usually 48 hours to 72hours)
  residual urine > 300ml diagnosed by bladder ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Jiwon Han, Ms, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Background] Hristovska AM, Duch P, Allingstrup M, Afshari A. Efficacy and safety of sugammadex versus neostigmine in reversing neuromuscular blockade in adults. Cochrane Database Syst Rev. 2017 Aug 14;8(8):CD012763. doi: 10.1002/14651858.CD012763. PMID 28806470